CLINICAL TRIAL: NCT02779803
Title: STAMCAR: A Prospective EC-IC Bypass Registry
Status: Withdrawn | Type: Observational
Why Stopped: The study team has made the decision to close this study at this time. No patient data was collected and/or analyzed. Since there was no study funds, contracts and budgets were unable to be drafted and sent to participating sites.
Sponsor: Lahey Clinic (Other)
Collaborators: American Association of Neurological Surgeons (Other)
Responsible Party: Sponsor
Other Study IDs: LCID: 2015-034
Record Dates: First submitted 2016-05-12; First posted 2016-05-20 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2021-08

CONDITIONS: Carotid Occlusion
MeSH Terms: interventions — Cerebral Revascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: EC-IC bypass — To determine if cerebral revascularization via STA to MCA bypass to improve cerebral hemodynamics, cognitive function, and quality of life in a defined subgroup of symptomatic carotid occlusion patients.

SUMMARY:
A prospective registry evaluating the efficacy of EC-IC bypass in a subgroup of patients, specifically, patients with carotid occlusion and symptoms refractory to medical therapy and evidence for poor cerebrovascular reserve as evaluated by physiological testing (e.g. Diamox Challenge SPECT Scan). This subgroup includes:

1. Hospitalized unstable patient with crescendo or postural TIA's
2. Patients with multiple TIA's, limb-shaking TIA's, and/or cognitive decline despite medical therapy.

DETAILED DESCRIPTION:
The registry is a multi-center international prospective registry. The patients will be prospectively followed for 24 months. Enrollment into the registry will take place over 3 years.

The primary objective is to collect prospective data on cerebral revascularization via superficial temporal artery (STA) to middle cerebral artery (MCA) for symptomatic carotid occlusion patients to determine if the procedure can be performed with less than 8% major peri-operative benchmark.

The secondary objective is to determine if cerebral revascularization via STA to MCA bypass will improve cerebral hemodynamics, cognitive function, and quality of life in a defined subgroup of symptomatic carotid occlusion patients over a 2 year period.

Clinical outcome in terms of resolved symptomatology, improved cerebrovascular hemodynamics, and cognitive status will be assessed. Short term and long term follow-up for a period of 24 months will include assessment of ipsilateral stroke or TIA rate, mortality, graft patency, assessment of MCA and bypass flow rates (if available), cognitive evaluation and quality of life evaluation.

Following enrollment baseline demographics and operative data will be collected. Follow-up will be performed at 1 month (m), 3m, 6m, 12m and 24m. Occurrence of new TIA or stroke will be determined. The patient's bypass patency, Qualitative Magnetic Resonance Angiogram (QMRA) flow data (site discretion) and NIHSS Score (NIHSS), Barthel Index (mBARTHEL), modified Rankin Scales (mRANKIN), EuroQOL, and the Montreal Cognitive Assessment (MoCA) with digital Clock Drawing (dCDT) will be recorded. An additional battery of neurocognitive tests will also be administered (Symbol Digit Modalities Test SDMT, Delis-Kaplan Executive Function System D-KEFS and TRAILS A/B).

ELIGIBILITY:
Inclusion Criteria:

* Internal carotid artery or middle cerebral artery occlusion
* Transient ischemic attack (TIA) or ischemic stroke in the ipsilateral hemisphere within 30 days in patients who are either

  * hospitalized unstable patients with crescendo or postural TIA's, OR
  * Multiple TIA's, limb-shaking TIA's, and/or cognitive decline despite medical therapy*
* Evidence of ipsilateral impaired cerebrovascular reserve on physiological testing (e.g. Diamox challenge SPECT)
* Modified Rankin Score (mRS) >3
* Language comprehension intact
* Age 18-85 years * failure of medical therapy must include at least failure on a regimen of antiplatelets and statins.

Exclusion Criteria:

* Moya-moya syndrome
* Known heart disease likely to cause cerebral ischemia

  * Prosthetic Valves
  * Atrial Fibrillation
  * Infective endocarditis
  * Left atrial or ventricular thrombus
  * Sick sinus syndrome
  * Cardiac myxoma
  * Cardiomyopathy with ejection fraction < 25%
* Any condition likely to lead to death within 2 years
* Pregnancy
* Allergy or contraindication to aspirin
* Uncontrolled diabetes mellitus (FBS > 300 mg%/16.7 mmol/L)
* Uncontrolled hypertension (systolic BP>180, diastolic BP >110), other than induced for control of pressure dependent symptoms
* Uncontrolled hypotension (diastolic BP <65)
* Unstable angina

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with internal carotid artery or middle cerebral artery occlusion and symptoms refractory to medical therapy and evidence for poor cerebrovascular reserve as evaluated by physiological testing (e.g. Diamox Challenge SPECT Scan).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Ipsilateral Ischemic Stroke | During surgery
Number of Patients with Ipsilateral Ischemic Stroke | Up to 30 days from surgery
Number of Patients that experience Stroke | After 30 days from surgery
Number of Patients that experience Death | After 30 days from surgery

SECONDARY OUTCOMES:
Cerebral Hemodynamic Testing | baseline, 3 months, 12 months
  Steal, Reduced reserve, normal (specific modality to be determined by site)
Qualitative Magnetic Resonance Angiogram, Non-invasive Optimal Vessel Analysis Blood Flow Data | baseline, 3 months, 12 months
  Site discretion; test assess the blood flow to the vessels in the brain
Bypass Patency | 3 months, 6 months, 12 months, 24 months
  Blood flow remains normal through the bypass
EuroQOL-5 Dimensions | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  A standardized instrument for use as a measure of health outcomes and is applicable to a wide range of health conditions and treatments; provides a simple description profile and a single index value for health status.
Montreal Cognitive Assessment (MoCA) | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  The MoCA was designated as a rapid screening instrument for mild cognitive dysfunction; it assesses difference cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
National Institutes of Health Stroke Scale (NIHSS) | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  A systematic assessment tool that provides a quantitative measure of stroke-related neurological deficit; used to evaluate acuity of stroke patients, determine appropriate treatment, and predict patient outcomes.
Modified Rankin Scale (mRankin) | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  A 6(0-5) point disability scale that is used widely in both secondary prevention and acute stroke trials, including most of the thrombolysis trials that ranks the patient based upon the disability symptoms
Modified Barthel Index (mBarthel) | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  The Barthel Index consists of 10 items that measure a person's daily functioning, specifically the activities of daily living and mobility. The items include feeding, moving from wheelchair to bed and return, grooming, transferring to and from a toilet, bathing, walking on level surface, going up and down stairs, dressing, continence of bowels and bladder. Can be used to monitor improvement in activities of daily living over time.
Digital Clock Drawing Test (dCDT) | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  The dCDT provides a novel technique to assess both cognitive and motor aspects of psychomotor speed within the same task and the potential to uncover subtleties of behavior not previously detected with non-digitized modes of data collection.
Delis-Kaplan Executive Function System (D-KEFS) | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  the D-KEFS Verbal Fluency Tests comprises of three testing conditions: Letter Fluency, Category Fluency, and Category Switching. This test measures the examinee's ability to generate words fluently in an effortful, phonetic format (Letter Fluency), from overlearned concepts (Category Fluency), and while simultaneously shifting between overlearned concepts (Category Switching).
Reitan Trails A/B Test | baseline, 1 month, 3 months, 6 months, 12 months, 24 months
  Cognitive Assessment; assess the examinee's ability visual attention and task switching abilities; the trails should be made quickly as possible while trying to avoid mistakes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos David, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Lahey Hospital & Medical Center, Burlington, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided